CLINICAL TRIAL: NCT03167840
Title: Falls Prevention Through Physical And Cognitive Training (Falls PACT) in Older Adults With Mild Cognitive Impairment: A Randomised Controlled Trial
Brief Title: Falls Prevention Through Physical And Cognitive Training in Mild Cognitive Impairment
Acronym: FallsPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Santo Tomas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20170402001
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2017-05

CONDITIONS: Mild Cognitive Impairment
Keywords: falls prevention, older adults, mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Restraint, Physical; Cognitive Training; Exercise; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical training alone (PT) (Experimental): Physical Training (flexibility, endurance, strengthening, and balance training) for 60-90 minutes 3x/week over 12 weeks of moderate intensity.
  Interventions: Behavioral: Physical Training
- Cognitive training alone (CT) (Experimental): Cognitive training with a focus on orientation, memory, attention and executive functioning for 60-90 minutes per session, once per week for 12 weeks.
  Interventions: Behavioral: Cognitive training
- Physical and cognitive training (PACT) (Experimental): Integrated cognitive training in physical exercise for 60-90 minutes per session, 3x/week over 12 weeks.
  Interventions: Behavioral: Physical and Cognitive Training
- Wait-list group (WG) (No Intervention): The control group on wait-list. They will be instructed to go on with their usual activities and will receive the intervention, combined physical and cognitive training, at a later date.

INTERVENTIONS:
Behavioral: Physical and Cognitive Training — Physical Exercise and Cognitive Training
  Other Names: Integrated cognitive training in physical exercise
  Arms: Physical and cognitive training (PACT)
Behavioral: Physical Training — Physical training alone
  Other Names: Physical exercise
  Arms: Physical training alone (PT)
Behavioral: Cognitive training — Cognitive training alone
  Other Names: Mental exercise
  Arms: Cognitive training alone (CT)

SUMMARY:
This randomised controlled trial aims to determine the effectiveness of combined physical and cognitive training in preventing falls and decreasing risks of falls among community-dwelling older persons with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
This is a single-blind, multicentre, randomised controlled trial. Community-dwelling older adults with MCI aged 60 or above will be recruited. They will be randomly allocated into four groups: Physical Training alone (PT), Cognitive Training alone (CT), combined Physical And Cognitive Training (PACT) and wait-list group (WG). Assessors blinded to participant allocation will conduct pre-test, posttest, and 6-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or above
* community-dwelling in Manila, Philippines
* diagnosed with MCI

Exclusion Criteria:

* diagnosis of dementia or Alzheimer's disease
* history of major medical conditions such as cerebrovascular disease, cardiopulmonary condition, serious musculoskeletal disease, cancer, major psychiatric condition
* have severe visual and/or hearing impairment
* taking medications such sedatives, antidepressants, diuretics, anti-epilepsy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Falls Rate | 9 months
  Number of Falls over a period of time

SECONDARY OUTCOMES:
Change in Physiologic Profile Assessment (PPA) score | Baseline, 3 months, 9 months
  Physiologic risk for falls
Change in Falls Risks for Older People in the Community (FROP-Com) Screen score | Baseline, 3 months, 9 months
  Overall fall risk
Change in Global Cognitive Function | Baseline, 3 months, 9 months
  Montreal Cognitive Assessment (MoCA)
Change in Memory Function | Baseline, 3 months, 9 months
  Memory Index Score of the Montreal Cognitive Assessment (MoCA-MIS)
Change in Executive Function | Baseline, 3 months, 9 months
  Executive Function Performance Test (EFPT)
Change in Balance | Baseline, 3 months, 9 months
  Time Up and Go Test (TUGT)
Change in Gait Speed | Baseline, 3 months, 9 months
  10-Meter Walk Test (10MWT)
Change in Muscle Strength | Baseline, 3 months, 9 months
  30s-Chair-Stand Test (CST)

OTHER OUTCOMES:
Change in Fear of Falling | Baseline, 3 months, 9 months
  Falls Efficacy Scale - International
Change in Quality of Life | Baseline, 3 months, 9 months
  European Quality of life - five dimensions - five levels (EQ-5D-5L) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: William Tsang, PhD, Principal Investigator — The Hong Kong Polytechnic University - Department of Rehabilitation Sciences
Locations (1):
- University of Santo Tomas, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lipardo DS, Tsang WWN. Falls prevention through physical and cognitive training (falls PACT) in older adults with mild cognitive impairment: a randomized controlled trial protocol. BMC Geriatr. 2018 Aug 24;18(1):193. doi: 10.1186/s12877-018-0868-2. PMID 30143002